CLINICAL TRIAL: NCT00957242
Title: AntiCoagulant Effectiveness in Idiopathic Pulmonary Fibrosis (ACE-IPF)
Brief Title: AntiCoagulant Effectiveness in Idiopathic Pulmonary Fibrosis
Acronym: ACE-IPF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Excess of mortality in the treatment group created safety concerns.
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00017156; 5U10HL080413-05 (NIH); 671
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2013-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; Warfarin
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- warfarin (Active Comparator): Oral warfarin titrated to an international normalization ratio (INR) of 2-3
  Interventions: Drug: warfarin
- placebo (Placebo Comparator): Oral placebo (1mg or 2.5mg)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: warfarin — Oral warfarin (1mg or 2.5mg) titrated to an INR of 2-3.
  Other Names: warfarin sodium
  Arms: warfarin
Drug: placebo — Oral placebo (1mg or 2.5mg)
  Arms: placebo

SUMMARY:
This study will test the effectiveness of warfarin in patients with IPF. Approximately 256 patients will be randomized 1:1 to either warfarin or placebo. Patients will return at week 1 for a safety review and every 16 weeks for 48 weeks. The primary endpoint in the study is the time to either death, non-bleeding/non-elective hospitalization, or a drop of greater than 10% in forced vital capacity (FVC) from baseline.

DETAILED DESCRIPTION:
Study design:

ACE-IPF was a double-blind, randomized, placebo-controlled trial of an oral warfarin dose adjusted to an international normalized ratio (INR) response of 2.0 to 3.0, compared with a sham dose-adjusted placebo. The trial was originally designed as an event-driven study with a treatment period of up to 144 weeks. Given the slow rate of recruitment and higher than anticipated event rates seen in another Idiopathic Pulmonary Fibrosis Clinical Research Network (IPFnet) trial, the protocol was modified to have a maximum treatment period of 48 weeks after eleven patients were enrolled in the study. Participants were to be seen at screening, baseline, and at 16, 32, and 48 weeks after enrollment.

Outcome measures:

The primary outcome was a composite endpoint based on the time to all-cause mortality; non-elective, non-bleeding hospitalization; or a decrease in the absolute FVC ≥10% from baseline value. Secondary outcome measures included rates of mortality, hospitalization, respiratory-related hospitalization, acute exacerbation, bleeding, cardiovascular events, and changes over time in FVC, six-minute walk test distance, diffusing capacity of lung for carbon monoxide (DLCO), plasma fibrin D-dimer levels, and quality of life (QOL) assessments.

Data Analysis Continuous variables at baseline were expressed as means (standard deviations) and medians (25th and 75th percentiles). Categorical variables at baseline were expressed as counts and percentages. Unadjusted estimates of event rates for time-to-event variables were computed using the Kaplan-Meier estimator with comparisons based on the log-rank test statistic. The primary hypothesis was tested using a Cox proportional hazards regression model, comparing the treatment effect on the primary composite endpoint. Pre-specified covariates in this model included an indicator variable for the treatment group and the DLCO measurement from the baseline assessment.

Randomization:

Subjects were randomly assigned to study arms in a 1:1 ratio, using a permuted-block design with varying block sizes, to receive either warfarin or matched placebo. Subjects were stratified by clinical center and a DLCO threshold of 35% of predicted. Randomization lists were generated by the study data coordinating center (DCC) and provided to a phone- and web-enabled registration system (Almac Clinical Services, Inc.) that allowed sites to enroll subjects and receive study kits while keeping the study team and subjects blinded to treatment assignment.

INR testing and monitoring:

Study subjects were provided two strengths of warfarin tablets (1 mg and 2.5 mg) or matching placebos. Subjects measured their INR with encrypted meters (INRatio®, Alere, San Diego, CA) at least weekly. Home monitoring was validated by plasma INR measurement at the week 1 and 16 visits. Individual INR meters and test strips were replaced and subjects were reinstructed if meter INR readings varied by more than 30% from the laboratory INR. Efficacy of home INR measures were determined by time-in-target INR range of all patients, calculated on the basis of linear interpolation, 12 after excluding readings taken at baseline, during initial warfarin titration (until INR ≥ 2.0), study drug interruption, or following the discontinuation of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF
* Age between 35 and 80, inclusive
* Capable of understanding and signing consent
* Progression despite conventional therapy (standard of care). Progression defined as:

  1. Worsened dyspnea
  2. FVC decreased by >=10% predicted OR
  3. DLCO decreased by >=10% absolute OR
  4. Reduction of oxygenation saturation >= 5% with or without exertion on a constant oxygen (02) administration
  5. Worsened radiographic findings (chest x-ray or high-resolution computed tomography)

Exclusion Criteria:

* Current enrollment in another investigational protocol
* Current treatment with an investigational drug (i.e., participating in an active investigational drug protocol) within the previous 4 weeks or 5 times the half-life of the investigational agent, whichever is longer, prior to screening
* Subject is actively listed for lung transplantation at the time of enrollment
* Subjects who will not be able to perform/complete the study, in the judgment of the physician investigator or coordinator, for at least 3 months. For example:

  1. Subject has current signs or symptoms of severe, progressive or uncontrolled comorbid illnesses such as: renal, hepatic, hematologic, gastrointestinal, endocrine, cardiac, neurologic, or cerebral disease, or any laboratory abnormality which would pose/suggest a risk to the subject during participation in the study.
  2. Subject has a transplanted organ requiring immunosuppression
  3. History of substance abuse (drugs or alcohol) within the 2 years prior to screening, history of noncompliance to medical regimens, inability or unwillingness to perform INR monitoring, or other condition/circumstance that could interfere with the subject's adherence to protocol requirements (e.g. psychiatric disease, lack of motivation, travel, etc).
  4. Have any known active malignancy or have a history of malignancy within the previous 2 years (an example of an exception is a non-melanoma skin cancer that has been treated with no evidence of recurrence for at least 3 months) that might increase the risk of bleeding.
* Estimated life expectancy < 12 months due to a non-pulmonary cause.
* Subject has another respiratory disease that is predominant (as judged by the PI) in addition to IPF.
* Anticoagulation-related exclusions include:

  1. Current anticoagulation therapy with warfarin
  2. Increased risk of bleeding (e.g. uncorrectable inherited or acquired bleeding disorder)
  3. Platelet count < 100,000 or hematocrit < 30% or > 55%
  4. History of severe gastrointestinal bleeding within 6 months of screening
  5. History of cerebral vascular accident (CVA) within 6 months of screening
  6. High risks of falls as judged by the PI
  7. Surgery or major trauma within the past 30 days
  8. Pregnancy, or lack of use of birth control method in women of childbearing age
  9. Any condition that, in the determination of the PI, is likely to require anticoagulation therapy during the study.
  10. Clopidogrel and aspirin combination therapy for > 30 days duration is exclusionary.

      (Aspirin monotherapy [81-325 mg daily] or clopidogrel monotherapy are acceptable. Combination clopidogrel and aspirin <=81mg/day for ≤30 days is also acceptable. NSAIDS are discouraged; acetaminophen may be substituted.)
  11. Patients on prasugrel are excluded. Prasugrel must be stopped for one week prior to starting study drug.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galen Toews, MD, Study Chair — University of Michigan; Gail Weinmann, MD, Study Director — National Heart, Lung, and Blood Institute (NHLBI); Kevin Brown, MD, Principal Investigator — National Jewish Health; Rob Kaner, MD, Principal Investigator — Weill Medical College at Cornell University; Talmadge King, MD, Principal Investigator — University of California, San Francisco; Joe Lasky, MD, Principal Investigator — Tulane University School of Medicine; James Loyd, MD, Principal Investigator — Vanderbilt University; Fernando Martinez, MD, Principal Investigator — University of Michigan; Imre Noth, MD, Principal Investigator — University of Chicago; Ganesh Raghu, MD, Principal Investigator — University of Washington; Jesse Roman, MD, Principal Investigator — Emory University; Jay Ryu, MD, Principal Investigator — Mayo Clinic; Joseph Lynch, MD, Principal Investigator — University of California, Los Angeles; Kevin Anstrom, PhD, Principal Investigator — Duke University; Joao deAndrade, MD, Principal Investigator — University of Alabama at Birmingham; Jeffrey Chapman, MD, Principal Investigator — The Cleveland Clinic; Lake Morrison, MD, Principal Investigator — Duke University; Michael Kallay, MD, Principal Investigator — Highland Hospital; Steven Sahn, MD, Principal Investigator — Medical University of South Carolina; Marilyn Glassberg, MD, Principal Investigator — University of Miami; Milton Rossman, MD, Principal Investigator — University of Pennsylvania; John Fitzgerald, MD, Principal Investigator — University of Texas; Mary Beth Scholand, MD, Principal Investigator — University of Utah; Neil Ettinger, MD, Principal Investigator — St. Luke's Hospital; Danielle Antin-Ozerkis, MD, Principal Investigator — Yale University
Locations (22):
- United States (22):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - Highland Hospital - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah Health Research Center, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625
- [Derived] Andrade J, Schwarz M, Collard HR, Gentry-Bumpass T, Colby T, Lynch D, Kaner RJ; IPFnet Investigators. The Idiopathic Pulmonary Fibrosis Clinical Research Network (IPFnet): diagnostic and adjudication processes. Chest. 2015 Oct;148(4):1034-1042. doi: 10.1378/chest.14-2889. PMID 26111071
- [Derived] Durheim MT, Collard HR, Roberts RS, Brown KK, Flaherty KR, King TE Jr, Palmer SM, Raghu G, Snyder LD, Anstrom KJ, Martinez FJ; IPFnet investigators. Association of hospital admission and forced vital capacity endpoints with survival in patients with idiopathic pulmonary fibrosis: analysis of a pooled cohort from three clinical trials. Lancet Respir Med. 2015 May;3(5):388-96. doi: 10.1016/S2213-2600(15)00093-4. Epub 2015 Apr 15. PMID 25890798
- [Derived] Noth I, Anstrom KJ, Calvert SB, de Andrade J, Flaherty KR, Glazer C, Kaner RJ, Olman MA; Idiopathic Pulmonary Fibrosis Clinical Research Network (IPFnet). A placebo-controlled randomized trial of warfarin in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2012 Jul 1;186(1):88-95. doi: 10.1164/rccm.201202-0314OC. Epub 2012 May 3. PMID 22561965
- See also: IPFnet Web Site — http://ipfnet.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized at 25 U.S. sites in a 1:1 ratio to warfarin or matching placebo for a planned treatment period of 48 weeks. International normalized ratios (INR) were monitored using encrypted home point-of-care devices that allowed blinding of study therapy.
Groups:
- Placebo: Oral placebo (1mg or 2.5mg)
  placebo : Oral placebo (1mg or 2.5mg)
- Warfarin: Oral warfarin titrated to an INR of 2-3
  warfarin : Oral warfarin (1mg or 2.5mg) titrated to an INR of 2-3.
Period: Overall Study
Arm/Group | Placebo | Warfarin
Started | 73 | 72
Completed | 73 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Warfarin | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 22 | 53
  >=65 years | 42 | 50 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (7.4) | 67.3 (7.1) | 67 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 24 | 39
  Male | 58 | 48 | 106
Region of Enrollment [Number; unit: participants]
  United States | 73 | 72 | 145

OUTCOME MEASURES:

1. Primary Outcome: Death, Non-bleeding/Non-elective Hospitalization, or >10% Drop in Forced Vital Capacity
Description: Death, non-bleeding/non-elective hospitalization, or >10% drop in forced vital capacity.
Time Frame: Events up to 48 weeks
Population: All participants per intention-to-treat (ITT)
Measure: Number; unit: events
Groups:
- Placebo: matched placebo
- Warfarin: warfarin sodium titrated to an INR of 2.0-3.0
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 73 | 72
events | 17 | 23
Statistical Analysis 1: Comparison: Placebo vs Warfarin; The study was designed to have 90% power to detect a difference in 48-week event free rates of 70% for the warfarin group versus 50% for the placebo group. A total of at least 95 adjudicated primary endpoints were required to achieve 90% power with 2-sided, type I error rate of 0.05 and a 1:1 randomization ratio. These calculations yielded a requisite total sample size of 256; Test type: Superiority or Other; p = 0.27, Regression, Cox; Prespecified covariates in the model included an indicator variable for the treatment group and the DLCO measurement from the baseline assessment; Cox Proportional Hazard = 1.32, 95% CI 2-sided [0.70 to 2.47] — Warfarin vs. Placebo

2. Secondary Outcome: All Cause Mortality
Time Frame: maximum of 48 weeks
Population: All participants per intention-to-treat (ITT)
Measure: Number; unit: events
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 73 | 72
events | 3 | 14
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.005, Cox Proportional; Cox Proportional Hazard = 5.03, 95% CI 2-sided [1.44 to 17.54]

3. Secondary Outcome: Change in Forced Vital Capacity (FVC) From Baseline to 16 Weeks
Description: Week-16 change from Baseline
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 44 | 42
liters | -0.07 (0.21) | -0.01 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.083, Mixed Models Analysis; t-value = 0.08, 95% CI [-0.01 to 0.17]

4. Secondary Outcome: All-cause Hospitalizations
Time Frame: maximum 48 weeks
Measure: Number; unit: events
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 73 | 72
events | 11 | 20
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.054, Cox Proportional; Hazard Ratio (HR) = 2.06, 95% CI 2-sided [0.99 to 4.31]

5. Secondary Outcome: Bleeding Events
Time Frame: maximum of 48 weeks
Measure: Number; unit: events
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 73 | 72
events | 3 | 4
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.19, Cox Proportional; Hazard Ratio (HR) = 2.47, 95% CI 2-sided [0.64 to 9.56]

6. Secondary Outcome: Acute Exacerbations of Idiopathic Pulmonary Fibrosis (IPF)
Time Frame: maximum of 48 weeks
Measure: Number; unit: events
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 73 | 72
events | 2 | 6
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.35, Cox Proportional; Hazard Ratio (HR) = 2.25, 95% CI 2-sided [0.41 to 12.34]

7. Secondary Outcome: Respiratory-related Hospitalizations
Time Frame: maximum 48 weeks
Measure: Number; unit: events
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 73 | 72
events | 2 | 6
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.15, Cox Proportional; Hazard Ratio (HR) = 3.24, 95% CI 2-sided [0.65 to 16.10]

8. Secondary Outcome: Cardiovascular Mortality or Morbidity
Description: Measured at 48 Weeks
Time Frame: maximum of 48 weeks
Measure: Number; unit: events
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 73 | 72
events | 8 | 12
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.88, Cox Proportional; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.24 to 3.39]

9. Secondary Outcome: Change in 6-minute Walk Distance (6MWD)
Description: The 6MWD is a measure of exercise tolerance. Change in exercise tolerance is calculated at the latest time point (up to 48 weeks) minus the earliest time point (at baseline).
Time Frame: Change from baseline to last visit (maximum of 48 weeks)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 73 | 72
meters | -16.41 (41.31) | 8.68 (178.91)
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.7222, Mixed Models Analysis; t-value = 10.88, 95% CI 2-sided [-49.57 to 71.34]

10. Secondary Outcome: Total Score St. George's Respiratory Questionnaire (SGRQ)
Description: The SGRQ is a quality of life measurement used to assess respiratory well being with a 0*-100 range (*indicates better health--lower is better).
Time Frame: Week 16 Change from Baseline
Population: All participants per intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 41 | 41
score on a scale | 1.66 (11.28) | 3.24 (12.32)
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.27, Mixed Models Analysis; t-value = -1.78, 95% CI 2-sided [-7.04 to 3048]

11. Secondary Outcome: Change in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) From Baseline to 16 Weeks
Description: The DLCO measures the partial pressure difference between inspired and expired carbon monoxide.
Time Frame: Week 48 / Final Visit
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 54 | 52
mL/min/mmHg | -1.41 (2.55) | -1.34 (3.07)
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.957, Mixed Models Analysis; t-value = 0.05, 95% CI 2-sided [-1.67 to 1076]

12. Secondary Outcome: Fibrin D-dimer Change From Baseline to 16 Weeks
Description: Biomarker that measures biologic activities in patients as opposed to response.
Time Frame: maximum of 48 weeks
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Placebo | Warfarin
Number analyzed (Participants) | 35 | 27
mg/ml | .02 (0.20) | -.61 (1.26)
Statistical Analysis 1: Comparison: Placebo vs Warfarin; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; t-value = -0.48, 95% CI 2-sided [-0.84 to -0.12]

ADVERSE EVENTS:
Time Frame: Collected during study participation period plus 4 weeks from last dose of study agent. Maximum of 52 weeks. Mean collection period with study termination was 32 weeks.
Arm/Group | Placebo | Warfarin
Serious Adverse Events (participants affected / at risk) | 12/73 | 21/72
Other Adverse Events (participants affected / at risk) | 28/73 | 16/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=73) | Warfarin (N=72)
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haeamothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Cario-Respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=73) | Warfarin (N=72)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 3 (3)
Headache (Nervous system disorders) | 8 (10) | 3 (3)
Dizziness (Nervous system disorders) | 5 (7) | 3 (5)
Oedema Peripheral (General disorders) | 5 (5) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 4 (7) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No